CLINICAL TRIAL: NCT00831207
Title: Beta-2 Microglobulin and Serum Cytokines as Indicators of Antiretroviral Therapy Failure
Brief Title: Beta-2 Microglobulin and Serum Cytokines x HAART
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Faculdade de Medicina de Botucatu, UNESP, Botucatu, Brasil (Other)
Responsible Party: Ricardo Augusto Monteiro de Barros Almeida, Faculdade de Medicina de Botucatu, UNESP, Botucatu, Brasil
Other Study IDs: upeclin/HC/FMB-Unesp-19
Record Dates: First submitted 2008-12-26; First posted 2009-01-28 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: HIV Patients
Keywords: B-2 microglobulin; Serum cytokines; HIV-1; Resistance; HAART; Therapeutic failure; Genotyping.

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- G1: 15 HIV-1+ individuals, previously untreated or without HAART for at least six months and CD4+ < 350 cells/mm3.
- G2: 31 HIV-1+ individuals undergoing HAART without virological therapeutic failure (TF).
- G3: 43 HIV-1+ individuals undergoing HAART with TF.
- G4: 20 normal individuals who served as controls for serum cytokines.

SUMMARY:
Cross-sectional study to assess the behavior of Beta-2 microglobulin and serum cytokines TNF-α, IFN-γ, IL-2, IL-4 and IL-10 as indicators of highly active antiretroviral therapy (HAART) failure.

DETAILED DESCRIPTION:
Objective: To assess the behavior of Beta-2 microglobulin and serum cytokines TNF-α, IFN-γ, IL-2, IL-4 and IL-10 as indicators of highly active antiretroviral therapy (HAART) failure Design: Cross-sectional study. Methods: Eighty-nine HIV-1+ patients and 20 normal individuals were divided into 4 groups: G1- 15 HIV-1+ individuals, previously untreated or without HAART for at least six months and CD4+ < 350 cells/mm3; G2- 31 HIV-1+ individuals undergoing HAART without virological therapeutic failure (TF), G3- 43 HIV-1+ individuals undergoing HAART with TF, and GC- 20 normal individuals who served as controls for serum cytokines. Demographic, clinical and HAART data were reviewed, and Beta-2 microglobulin, serum cytokines (TNF-α, IFN-γ, IL-2, IL-4 and IL-10), HIV-1 genotyping, plasma viral load and CD4+ and CD8+ lymphocytes tests were performed.

Key words: Beta-2 microglobulin, serum cytokines, HIV-1, resistance, HAART, therapeutic failure, genotyping.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1-infected individuals
* Over 18 years old
* Sign the "written consent form" (WCF)

Exclusion Criteria:

* Do not presenting other immunosuppression causes, such as neoplasias, transplantations
* Do not presenting treatment by immunosuppressive substances
* Do not presenting auto-immune diseases
* Not be using any type of immunostimulating substances
* Not at any time of gestation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 89 HIV-1-infected individuals assisted by the Tropical Diseases Sector of the Botucatu School of Medicine - UNESP and 20 normal blood donors at the Botucatu Blood Bank.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2004-08; Primary Completion 2005-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To assess the behavior of Beta-2 microglobulin as indicator of highly active antiretroviral therapy (HAART) failure. | At subject enrollment.

SECONDARY OUTCOMES:
To assess the behavior of serum cytokines TNF-α, IFN-γ, IL-2, IL-4 and IL-10 as indicators of highly active antiretroviral therapy (HAART) failure. | At subject enrollment.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo MB Almeida, MSc, Principal Investigator — Departamento de Doencas Tropicais e Diagnostico por Imagem - Faculdade de Medicina de Botucatu - UNESP.
Locations (1):
- Faculdade de Medicina de Botucatu - UNESP, Botucatu, São Paulo, Brazil